CLINICAL TRIAL: NCT02383797
Title: Immunodeficiency in Cartilage-hair Hypoplasia: Correlation With Pulmonary Disease, Infections and Malignancy
Brief Title: Immunodeficiency in Cartilage-hair Hypoplasia: Sub-project on Safety of Vaccination Against Chickenpox
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paula Klemetti, MD, PhD, Consultant in pediatric gastroenterology and immunology, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TYH2013336
Record Dates: First submitted 2015-02-10; First posted 2015-03-09 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Cartilage-hair Hypoplasia
MeSH Terms: conditions — Cartilage-hair hypoplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cartilage-hair hypoplasia (CHH) (Experimental): Selected CHH patients will be vaccinated against varicella with Varilrix, one dose of 0,5 ml subcutaneously. If no response is documented to the first dose, the second dose of 0,5 ml can be administered.
  Interventions: Biological: Varilrix

INTERVENTIONS:
Biological: Varilrix — Vaccination against varicella in selected cartilage-hair hypoplasia patients
  Other Names: ATC J07BK01

SUMMARY:
The investigatoris will carefully select cartilage-hair hypoplasia patients unexposed to varicella (VZV) and immunize patients in a controlled manner with VZV vaccine. Patients will be selected on the basis of disease severity and the degree of immunodeficiency (including CD4+ T-cell counts). Any potential complication of VZV immunization, such as rash, will be discussed with the patients/caregivers beforehand and acyclovir will be used to treat any VZV related symptoms, consistent with the current practices. The investigators will verify the development of immune response to vaccination by testing for VZV antibodies and cell-mediated immunity.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed cartilage-hair hypoplasia diagnosis
* age >12 months
* no history of chickenpox
* informed concent of the patient/caregiver.

Exclusion Criteria:

* positive serum IgG for varicella zoster virus
* low CD4+ cell counts (<15% or <200 cells/mm3)
* clinical or laboratory signs of severe immunodeficiency
* ongoing intravenous or subcutaneous immunoglobulin treatment

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2019-10 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Humoral response to vaccination | 4-6 weeks post-vaccination
Cell-mediated response to vaccination | 4-6 wks post-vaccination
Number and severity of adverse events to vaccination | 0-60 days

CONTACTS AND LOCATIONS:
Overall Officials: Outi Mäkitie, PhD, Study Director — Helsinki University Central Hospital and University of Helsinki, Folkhälsan Research Centre, Helsinki Finland

REFERENCES:
- [Derived] Vakkilainen S, Kleino I, Honkanen J, Salo H, Kainulainen L, Grasbeck M, Kekalainen E, Makitie O, Klemetti P. The Safety and Efficacy of Live Viral Vaccines in Patients With Cartilage-Hair Hypoplasia. Front Immunol. 2020 Aug 11;11:2020. doi: 10.3389/fimmu.2020.02020. eCollection 2020. PMID 32849667